CLINICAL TRIAL: NCT02550444
Title: Comparison Between Intravenous and Intrathecal Clonidine in Post-cesarean Analgesia
Brief Title: Intrathecal Clonidine in Cesarean Section May Lead to Worse Blood Gas Results in the Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE 05847312.8.0000.0068
Record Dates: First submitted 2015-09-04; First posted 2015-09-15 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2015-09

CONDITIONS: Pregnancy
Keywords: Clonidine; Anesthesia, Obstetrical
MeSH Terms: interventions — Clonidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Intravenous and intrathecal Placebo (Saline 0,9%); Intrathecal heavy Bupivacaine 0,5% (15mg), morphine 0,02 (80mcg) and fentanyl (10mcg).
  Interventions: Drug: Placebo
- Intrathecal Clonidine (Experimental): Intrathecal Adjuvant Clonidine 75 mcg; Intravenous Placebo (Saline 0,9%); Intrathecal heavy Bupivacaine 0,5% (15mg), morphine 0,02 (80mcg) and fentanyl (10mcg).
  Interventions: Drug: Intrathecal Clonidine
- Intravenous Clonidine (Experimental): Intravenous Clonidine 75 mcg; Intrathecal Placebo (Saline 0,9%); Intrathecal heavy Bupivacaine 0,5% (15mg), morphine 0,02 (80mcg) and fentanyl (10mcg).
  Interventions: Drug: Intravenous Clonidine

INTERVENTIONS:
Drug: Intrathecal Clonidine — Intrathecal Adjuvant Clonidine 75 mcg; Intravenous Placebo (Saline 0,9%); Intrathecal heavy Bupivacaine 0,5% (15mg), morphine 0,02 (80mcg) and fentanyl (10mcg).
  Other Names: Clonidine
  Arms: Intrathecal Clonidine
Drug: Intravenous Clonidine — Intravenous Clonidine 75 mcg; Intrathecal Placebo (Saline 0,9%); Intrathecal heavy Bupivacaine 0,5% (15mg), morphine 0,02 (80mcg) and fentanyl (10mcg).
  Other Names: Clonidine
  Arms: Intravenous Clonidine
Drug: Placebo — Intravenous and intrathecal Placebo (Saline 0,9%); Intrathecal heavy Bupivacaine 0,5% (15mg), morphine 0,02 (80mcg) and fentanyl (10mcg).
  Other Names: Saline
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate effects of intravenous clonidine in acute and chronic post-cesarean pain, possible adverse effects over mother-newborn pair, in comparison to intrathecal adjuvant clonidine and placebo.

DETAILED DESCRIPTION:
METHODS Patients The research was submitted and approved by the Clinics Hospital of University of São Paulo Ethics in Research Board (CAAE 05847312.8.0000.0068, Nº 940.941). Patients authorized their participation and the proposed interventions and data collection, through signature of Free Consent Term.

Inclusion criteria were women aged 18 years or older, in term pregnancy, who underwent elective cesarean (no labor). Exclusion criteria was the following: multiple pregnancy; moderate or several systemic disease, categorized as American Society of Anesthesiology physical status (ASA) higher or equal to 3; contraindications for spinal anesthesia; contraindications for the drugs involved in the study; uncontrolled high blood pressure or diabetes mellitus in need of insulin therapy; intravenous psychotropic drugs users; previously known malformation on the fetus; and patients with previous history of chronic pain.

Patients anesthetic management All volunteers were managed according to the hospital protocol for cesarean delivery, and the one difference between groups was the clonidine or placebo given intrathecally or intravenously. Multiparameter non-invasive monitoring was used. The patients received a intravenous 10ml/kg Ringer Lactate bolus during realization of spinal anesthesia with heavy Bupivacaine 0,5% (15mg), morphine 0,02 (80mcg) and fentanyl (10mcg). Blood pressure was measured non-invasively during intra-operative period, each 1 minute until the baby was born, and each 3 minutes after the delivery. Low blood pressure was treated with Metaraminol 0,2mg intravenous bolus and/or Ephedrine 5mg intravenous bolus. Bradycardia was defined as heart rate inferior to 45 beats per minute, and treated with Atropine 0,5mg intravenous bolus. Intra-operative rescue analgesia was provided, if necessary, according to the patients needs or if the assistant anesthetist felt that it was necessary, with Fentanyl intravenous bolus, until a maximum dose of 100mcg. Before the skin incision, the patient received cefazolin 2g IV. After cord clamp, patients received Oxytocin 5 international units diluted in Ringer Lactate 250ml, ketoprofen 100mg IV, Dipyrone 2g IV, Omeprazole 40mg IV, Ondansetron 8mg IV. After procedure, the women were driven to Post Anesthetic Care Unit (PACU). There, if they felt pain, they could receive morphine 2mg IV, each 5 minutes, according to the patients needs. Post-operative pain control in the ward was standardized on the following protocol: ketoprofen 100mg IV 12/12h, Dipyrone 2g IV 6/6h; Tramadol IV 100mg maximum 8/8h, if uncontrolled pain. If pain persists, morphine subcutaneously, 5mg could be administered by nurse, 4/4h. Nauseas were treated with Dimenhydrinate 50mg IV 6/6h and Metoclopramide 10mg IV 8/8h, and itch was attenuated with Diphenhydramine 25mg IV, in case of such symptoms.

A neonatology team was present in every delivery and was responsible for the first evaluation of the newborn, including Apgar score and resuscitation.

Groups and interventions The included patients were randomly divided into one of three groups. The professional who administered the drugs was external to de research group, and did it unblinded. The researcher who did the assessments of the variables was blind for what intervention had been made. In control group, patients received placebo intravenously and intrathecally. In the intrathecal clonidine group, patients received 75 mcg of spinal clonidine, and intravenous placebo. In the intravenous clonidine group, patients received 75 mcg of intravenous clonidine, and spinal placebo. The solutions volumes were the same in all three groups, by 0,9% saline fluid addition to intrathecal and intravenous infusions.

Outcomes Data including age, height, weight, body mass index (BMI), number of pregnancies, number of deliveries, associated morbidities, American Society of Anesthesiology (ASA) physical status classification, reason to cesarean, length of anesthesia, amount of fluids needed, basal blood pressure, minimum and maximum values, heart rate variation, vasopressor and chronotropic drugs need, anesthesia complications, adverse effects (nauseas, vomits, itch and shivering) and analgesic complementation intra-operative needs were registered. Systolic, diastolic and mean hypotension was considered when values decreased more than 20% of basal values. During the stay at PACU, motor block duration (time from beginning of the anesthesia until the patient be able to do 90º flexion movement of tights over hips and 90º flexion movement of legs over tights, on both inferior limbs, simultaneously and sustained for 5 seconds or more), pain and adverse effects were evaluated. Patients were assessed by researchers in 6, 12, 24 and 48 hours after spinal anesthesia induction. Post-operative pain was measured using a number verbal scale (NVS), from 0 to 10 (0 is equivalent to no pain at all and 10 means the worst pain ever). Patients informed their pain in rest and after been asked to change from the lying position to the sitting position. Treatment satisfaction was evaluated using a 0-10 scale, in which 0 meant unsatisfied and 10 full satisfaction. Patients were asked by research team to quantify the intensity of itch, nausea, vomit and dizziness in a four points scale (0=none, 1=mild, 2=moderate, 3=severe). Sedation was measured by the Richmond Agitation and Sedation Scale.

After 3 months, the women were evaluated trough a individual telephone call by a member of study team, when they were asked if they had any pain or abnormal sensation (burning, itch and numbness) at the section site; if they had any functional limitation due to pain; if they needed any drug for section site pain in last week; if they were nursing; and if the not-nursing reason was due to pain.

Newborn data included gestational age, weight after born, Apgar score at first, fifty and tenth minutes, umbilical artery blood gas analysis, and Neonatal Intensive Care Unit (ICU) admission need.

ELIGIBILITY:
Inclusion Criteria:

* term pregnancy;
* elective cesarean (no labor).

Exclusion Criteria:

* multiple pregnancy;
* moderate or several systemic disease, categorized as American Society of Anesthesiology physical status (ASA) higher or equal to 3;
* contraindications for spinal anesthesia;
* contraindications for the drugs involved in the study;
* uncontrolled high blood pressure or diabetes mellitus in need of insulin therapy;
* intravenous psychotropic drugs users;
* previously known malformation on the fetus;
* patients with previous history of chronic pain.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Umbilical Artery Blood Gas Analysis - pH | Right after born
  pH
Umbilical Artery Serum Lactate | Right after born
  Lactate
Newborn Apgar Score | First, Fifth and Tenth minutes after born
  Score can vary from 0 to 10.

SECONDARY OUTCOMES:
Maternal heart rate | Intraoperatively
  Heart rate during anesthesia
Maternal blood pressure variation | Intraoperatively
  Maximum and minimum blood pressure values
Numerical verbal scale for pain | 6, 12, 24 and 48 hours after cesarean section
  Score varies from 0 to 10
Maternal sedation | Intraoperatively
  Richmond Agitation and Sedation Scale (varies from -5 to +4)

CONTACTS AND LOCATIONS:
Overall Officials: Hermann S Fernandes, MD, Principal Investigator — Clinics Hospital of University of São Paulo Medical School

REFERENCES:
- [Background] Mayor S. 23% of babies in England are delivered by caesarean section. BMJ. 2005 Apr 9;330(7495):806. doi: 10.1136/bmj.330.7495.806-a. No abstract available. PMID 15817536
- [Background] Eisenach JC, De Kock M, Klimscha W. alpha(2)-adrenergic agonists for regional anesthesia. A clinical review of clonidine (1984-1995). Anesthesiology. 1996 Sep;85(3):655-74. doi: 10.1097/00000542-199609000-00026. No abstract available. PMID 8853097
- [Background] Filos KS, Goudas LC, Patroni O, Polyzou V. Intrathecal clonidine as a sole analgesic for pain relief after cesarean section. Anesthesiology. 1992 Aug;77(2):267-74. doi: 10.1097/00000542-199208000-00008. PMID 1642346
- [Derived] Fernandes HS, Bliacheriene F, Vago TM, Corregliano GT, Torres ML, Francisco RP, Ashmawi HA. Clonidine Effect on Pain After Cesarean Delivery: A Randomized Controlled Trial of Different Routes of Administration. Anesth Analg. 2018 Jul;127(1):165-170. doi: 10.1213/ANE.0000000000003319. PMID 29596102